CLINICAL TRIAL: NCT00953446
Title: Arterial Spin Labeling Blood Flow Magnetic Resonance Imaging for the Evaluation of the Response to Therapy With the Combination of Sunitinib and AMG386 in Metastatic Renal Cell Carcinoma
Brief Title: Arterial Spin Labeling Blood Flow Magnetic Resonance Imaging for the Evaluation of Response to Therapy in Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Amgen (Industry)
Responsible Party: Sponsor
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-105
Record Dates: First submitted 2009-08-05; First posted 2009-08-06 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Renal Cell Carcinoma
Keywords: metastatic renal cell carcinoma; ASL MRI; sunitinib; AMG386
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arterial Spin Labeling Blood Flow Magnetic Resonance Imaging (Experimental): * ASL MRI
  * Performed at baseline, 2 weeks upon initiation of therapy, after cycle 2 and/or cycle 4 of therapy, and at the end of treatment
  Interventions: Procedure: Arterial Spin Labeling Blood Flow Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Arterial Spin Labeling Blood Flow Magnetic Resonance Imaging — Performed at baseline, 2 weeks upon initiation of therapy, after cycle 2 and/or cycle 4 of therapy, and at the end of treatment
  Other Names: ASL MRI

SUMMARY:
The purpose of this study is to assess magnetic resonance imaging (MRI) as a tool to track tumor growth for renal cell carcinoma while participants are on clinical treatment therapy of sunitinib and AMG386. An MRI is a type of scan that uses powerful magnets to make clearer images or to focus on detailed medical information in the abdomen and pelvis. The imaging done for this study will use the arterial spin labeling (ASL) MRI technique that allows us to see blood flow changes which possibly may indicate changes in tumor growth. Participants will be on a clinical trial for the treatment.

DETAILED DESCRIPTION:
All participants must be enrolled on protocol, "Collection of Specimens and Clinical Data from Patients with Renal Cell Carcinoma Treatment with Targeted Therapies", about to start a treatment course with sunitinib and AMG386, and willing to come in for successive MRIs at the following times: baseline, 2 weeks upon initiation of therapy with sunitinib and AMG386, after cycle 2 and/or cycle 4 of therapy, and at the end of your study therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Patients diagnosed with metastatic renal cell carcinoma and who will initiate therapy with the combination of sunitinib and AMG386 as either their first anti-angiogenic therapy or after failure of prior cytokine therapy
* Enrolled on protocol 06-105, "Collection of specimens and clinical data from patients with renal cell carcinoma treated with targeted therapies"
* Found to have tumors that are >/=2.5 cm as determined by CT imaging
* Candidate lesions for ASL MRI should be >/= 2.5cm. Order of preference of lesion location will be as follows: abdominal lesions, bone lesions and chest lesions

Exclusion Criteria:

* Subjects will be excluded from the study if they have a contraindication to MRI which may include the following: Pacemaker, MRI incompatible metal implant, recently implanted vascular clip, history of claustrophobia, metal fragment within the eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-06-15 (Actual); Primary Completion 2011-09-13 (Actual); Study Completion 2011-09-13 (Actual)

PRIMARY OUTCOMES:
To explore the association of baseline blood flow in renal cell carcinoma(RCC) measured by ASL MRI and tumor response to treatment with the combination of sunitinib and AMG386 | 2 years
To explore the association of changes in tumor blood flow that occur early in the course of therapy compared to baseline and response of RCC to treatment with the combination of sunitinib and AMG386 | 2 years
To evaluate the association between changes in tumor blood flow on ASL over the course of therapy and at the time of disease progression and resistance to therapy. | 2 years
To compare above results to those observed in a comparable patient population receiving sunitinib alone. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Pedrosa, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts